CLINICAL TRIAL: NCT06930482
Title: Effect of SAFE Early Intervention Program on Neurodevelopmental Outcomes At 1 Year of Age in Infants at Risk of CP
Brief Title: Evaluation of The Effectiveness of The SAFE Early Intervention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayse Simsek, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 91610558-302.08.01-122723
Record Dates: First submitted 2025-04-01; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Preterm; Sensory Disorders; Cerebral Palsy
MeSH Terms: conditions — Premature Birth; Sensation Disorders; Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAFE Early Intervention Group (Experimental)
  Interventions: Behavioral: Safe early intervention; Behavioral: early intervention approach based on neurodevelopmental treatment
- Control Group (Other)
  Interventions: Behavioral: Safe early intervention; Behavioral: early intervention approach based on neurodevelopmental treatment

INTERVENTIONS:
Behavioral: Safe early intervention — The SAFE early intervention approach, an activity-focused, sensory intervention program, was applied to the babies in the intervention group in an enriched environment. As part of the intervention, coaching was provided in collaboration with the family on how to support the baby's development. For this purpose, family visits were made 15 days after the initial assessment and once a month. During these visits, the suggestions given to the family were repeated and all questions about the process were answered. It was discussed how the home environment should be structured in a way that is appropriate for the baby's development. The aims of the approaches applied were explained and information was provided about the follow-up process. In order to follow up on whether the family implemented the intervention, the family was interviewed by phone and the family was asked to keep an activity diary.
Behavioral: early intervention approach based on neurodevelopmental treatment — Within the scope of the study, NGT-based applications were applied to the babies included in the control group by their families. After the first assessment, activities were planned to support skills appropriate to the child's developmental level. The treatment movements, how to facilitate the baby's movements, and how to provide hand contact were demonstrated to the families in practice. The applicability of the intervention program was monitored with weekly phone calls. The babies were called to the clinic environment for a check-up every month to revise the intervention program and teach new movements, and an evaluation was made. Two home visits were made to evaluate the families' home environments and parental attitudes (pre- and post-intervention).

SUMMARY:
In this study, it was aimed to examine the effect of SAFE, which is a sensory-based, activity-oriented early intervention approach applied in an enriched environment with family cooperation, on cognitive, language, motor and sensory development in 3-6 months old risky infants. 46 infants with neurodevelopmental risk, whose corrected age was 3 months, were included in the study. Infants were randomly divided into two groups. Infants in the treatment group were included in an early intervention program according to the SAFE approach. Infants in the control group were included in the family education program based on the principles of Neurodevelopmental Therapy (NDT). The intervention was performed for 12 weeks, and all infants were evaluated with Bayley Developmental Scale for Infants and Young Children III (Bayley III) by a blinded investigator before treatment (3rd months) after treatment (6th months) and 12th months.

ELIGIBILITY:
Inclusion Criteria:• Corrected age of 3 months

* Any neurodevelopmental risk (perinatal stroke, perinatal asphyxia, HIE, GMK-IVK, PVL or gestational age of 32 and below)

Exclusion Criteria: • Having a congenital anomaly

* Having a genetic syndrome diagnosis (e.g. Down Syndrome)
* Parents do not speak Turkish

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Bayley Scales of Development for Infants and Toddlers III (Bayley-III) | 3 months,6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Yildiz R, Yildiz A, Apaydin U, Efkere PA, Gucuyener K, Hirfanoglu IM, Elbasan B. Long-Term Neurodevelopmental Outcomes of the SAFE Early Intervention in Infants at Risk: A Randomised Controlled Trial. J Paediatr Child Health. 2025 Oct;61(10):1662-1670. doi: 10.1111/jpc.70191. Epub 2025 Sep 2. PMID 40891629